CLINICAL TRIAL: NCT06787287
Title: A Study on the Application of Simple and Improved Radial Artery Compression Method After Transradial Coronary Intervention A Randomized, Controlled Clinical Trial
Brief Title: A Study on the Application of Simple and Improved Radial Artery Compression Method After Transradial Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guozhe Sun (Other)
Responsible Party: Sponsor-Investigator, Guozhe Sun, sub-investigator of Department of Cardiology in First Hospital of China Medical University, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 【2023】2023-341-2
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Radial Artery Occlusion
Keywords: percutaneous coronary intervention; Compression method; Radial artery complication
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The experimental group adopted improved compression method (Experimental): The experimental group adopted the improved compression method. A thick gauze block of 9cm*16cm*8mm was folded three times and placed at the puncture site of the patient's radial artery, and a spiral radial artery hemostatic device was placed above it. After rotating the hemostatic device several times clockwise to confirm that there was no bleeding at the puncture site, and then rotating the hemostatic device counterclockwise to make the radial artery hemorrhage occurred. The hemostatic device was turned clockwise again to stop the bleeding of the radial artery, and then turned counterclockwise every 1 hour. After continuous pressure on the puncture site for 4 hours, the band was removed and sterilized and covered with sterile dressing. Patients were monitored for at least 30 minutes after the band was removed. If the bleeding reappears, re-apply the band and repeat the process.
  24 hours after surgery, color Doppler ultrasound was used to determine the presence or absence of a radial
  Interventions: Procedure: Modified compression method
- The control group was treated with traditional compression method (No Intervention): The control group was treated with the traditional compression method. The spiral radial artery hemostatic device was applied at the radial artery puncture, and the radial artery was completely hemostatic after several turns clockwise, and then the radial artery was completely hemostatic after counterclockwise rotation, and then the radial artery was stopped bleeding after one turn clockwise rotation, that is, the minimal pressure was applied to ensure successful hemostasis. Then the hemostat was turned counterclockwise every 1 hour, and the puncture site was pressed continuously for 4 hours. The band was removed and covered with sterile dressing after disinfection. Patients were monitored for at least 30 minutes after the band was removed. If the bleeding reappears, re-apply the band and repeat the process.
  24 hours after surgery, color Doppler ultrasound was used to determine the presence or absence of a radial

INTERVENTIONS:
Procedure: Modified compression method — In the experimental group, an improved compression method was adopted. A thick gauze block of 9cm*16cm*8mm was folded three times and placed at the puncture site of the patient's radial artery, and a spiral radial artery hemostatic device was placed above it. The control group was treated with traditional compression method, and the spiral radial artery hemostat was applied directly at the radial artery puncture
  Arms: The experimental group adopted improved compression method

SUMMARY:
The objective of this study was to evaluate the specific effect of a simple modified method of thick gauze (9cm*16cm*8mm) combined with a hemostatic device in the prevention of early radial artery occlusion and other related vascular complications after transradial coronary intervention.

DETAILED DESCRIPTION:
Clinically, coronary intervention through radial artery is a common path for cardiovascular interventional therapy in recent years, and relevant clinical RCT studies and meta-analyses have confirmed that transradial intervention (TRI) has more benefits than transfemoral artery. Including reducing patient pain, easy pressure hemostasis, postoperative patients can not have to stay in bed, fewer vascular complications, reduce patient hospitalization costs and other advantages. However, radial artery occlusion (RAO) and hematoma are the most common postoperative complications of TRA. Although the vast majority of cases are asymptomatic from an ischemia perspective, it rules out ipsilateral TRA for future surgery. In particular, RAO will restrict the use of the radial artery to create an arteriovenous fistula for patients requiring hemodialysis, in addition to the fact that patients at high blood risk may not receive the benefits of the radial artery access in the case of repeat surgery. Therefore, the prevention of postoperative RAO is of fundamental clinical importance. Among the various strategies used to prevent RAO, postoperative arterial compression time and arterial compression level are important factors in changing the occurrence of RAO. In the CRASOC study, which included 3616 patients who were randomly divided into 3 groups, the incidence of RAO was 2.3% when hemostatic compression (10 ml of air) was light and short (1.5 hours). The incidence of RAO was 7.9% when hemostatic compression was lighter (10 ml of air) but longer (4 hours) and 9.4% when stronger pressure was applied (13 ml of air) and longer (4 hours), and the CRASOC trial highlights the effectiveness of combining a minimum pressure strategy with a short compression duration for the prevention of RAO. However, a very short compression duration may increase the rate of rebleeding at the puncture site, resulting in a renewed need for increased hemostatic pressure, which may paradoxically increase the incidence of RAO.

At present, when traditional pressure hemostasis is difficult in clinic or postoperative pressure pain is unbearable, our center often adopts a simple and improved method of thick gauze block (9cm*16cm*8mm) combined with hemostatic device, which can significantly improve the hemostatic effect. However, this method is only in the experience of single-center surgeons and has not been verified by relevant clinical studies. The center intends to conduct this clinical study to systematically evaluate the application effect of this improved compression method in radial artery compression hemostasis after transradial coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, regardless of gender;
* Patients undergoing coronary intervention;
* Patients with a transradial approach;
* Voluntarily participate and sign informed consent;

Exclusion Criteria:

* Intraoperative Allen test was positive for all patients;
* The intraoperative Barbeau tests were all D grade radial artery patients;
* Patients with blood or liver diseases;
* Patients with vascular diseases or malformations in the forearm;
* Patients with a history of RAO at baseline of the radial artery on the approach;
* Approach side arteriovenous fistula dialysis patients;
* Patients with subclavian artery occlusive disease (definite medical history or the difference in systolic blood pressure between the two upper limbs is more than 20mmHg);
* Patients who have completed coronary intervention (full heparin);
* Active bleeding at the puncture site before extraction;
* Systolic blood pressure greater than 180 mm Hg or diastolic blood pressure greater than 110 mm Hg at closure;
* Pregnant women or patients who are trying to conceive and have family plans;
* Patients whom the investigator deems inappropriate to participate in the clinical trial;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1568 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Incidence of 24-hours RAO (radial artery occlusion) | Acute radial artery occlusion was evaluated at 24 hours after the percutaneous coronary intervention
  Color Doppler ultrasound was used to determine the incidence of RAO (radial artery occlusion) at 24 hours after the percutaneous coronary intervention in both groups

SECONDARY OUTCOMES:
Occurrence of forearm hematomas | Within 24 hours after the procedure
  Forearm hematomas were recorded and graded using the EASY (Early Discharge After Transradial Stenting of Coronary Arteries) classification system, based on size and clinical presentation.
Postoperative pain within 24 hours | 24 hours after the procedure
  Pain intensity at the puncture site was assessed using the Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain).
Presence of palm swelling | Within 24 hours after the procedure
  Palm swelling was defined as a circumference increase of more than 0.5 cm compared with baseline, measured at the same palm location using a flexible tape measure.
Occurrence of forearm cyanosis | Within 24 hours after the procedure
  Cyanosis was visually assessed and defined as discoloration (bluish or purple tint) of the forearm skin, indicating impaired circulation.
Presence of finger numbness | Within 24 hours after the procedure
  Numbness was assessed by patient report and physical examination, defined as subjective loss or reduction of sensation in one or more fingers on the puncture side.
Incidence of tension blisters at the puncture site | Within 24 hours after the procedure
  Tension blisters were visually assessed and categorized as mild (small, localized, minimal pain) or severe (large, spreading, or with associated significant pain), based on extent and patient-reported symptoms.
Change in radial artery diameter from baseline | From baseline to 24 hours post-procedure
  Radial artery internal diameter was measured using color Doppler ultrasound at baseline and at 24 hours after the procedure, and the change was calculated to assess vascular response.

CONTACTS AND LOCATIONS:
Overall Officials: Yingxian Sun, Principal Investigator — First Hospital of China Medical University
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China